CLINICAL TRIAL: NCT01047878
Title: Genomic Analysis of Pediatric Bone Tumors (Other Title: Pediatric Bone Tumor Biology Study)
Brief Title: Genomic Analysis of Pediatric Bone Tumors
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: PEDSSARC0001; 97630 (Other: Stanford University Alternate IRB Approval Number); SU-12082009-4522 (Other: Stanford University)
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Bone Cancer
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor samples and blood

SUMMARY:
To determine whether gene expression analysis of primary tumor samples before and after chemotherapy are predictive of long-term survival in pediatric patients with bone sarcomas (Ewings sarcoma (ES) and Osteosarcoma(OS)).

ELIGIBILITY:
Inclusion Criteria:All patients with bone x-rays suggestive of a malignant bone tumor Exclusion Criteria:Patients with a known diagnosis of cancer.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients with bone x-rays suggestive of a malignant bone tumor
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2007-08; Primary Completion 2018-06 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
% necrosis post chemotherapy | his is measured at the time of sample collection since we are looking for % necrosis in the sample we are collecting
overall survival and event free survival | This is measured at the time the patient dies, or at the time when patient relapses from their disease. There is no set time since this outcome is individually assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Arun A Rangaswami, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States